CLINICAL TRIAL: NCT06225453
Title: Effect of Individualized Versus Conventional Blood Pressure Management on Major Adverse Cardiac, Cerebrovascular, and Renal Events After Major Non-cardiac Surgery: Multicenter, Randomized Controlled Trial
Brief Title: Individualized Versus Conventional Perioperative Blood Pressure Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Karam Nam, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPROUT-4
Record Dates: First submitted 2024-01-08; First posted 2024-01-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Major Non-cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized strategy (Experimental): Targeting mean arterial pressure and systolic blood pressure of ≥ -20% of their baseline values in each patient during surgery. The baseline values are defined as the average of all measurements between one day before surgery and the morning of the surgery. The target is applied until discharge from the post-anesthesia care unit. If the patient is transported to the intensive care unit after surgery, not the post-anesthesia care unit, then the strategy is applied until the end of surgery.
  The target is applied until discharge from the post-anesthesia care unit. It the patient is transported to the intensive care unit after surgery, not the post-anesthesia care unit, then the strategy is applied until the end of surgery.
  Interventions: Other: Individualized perioperative blood pressure management strategy
- Conventional strategy (Active Comparator): Targeting a mean arterial pressure of 65 mmHg or higher and a systolic blood pressure of 90 mmHg or higher during surgery. The target is applied until discharge from the post-anesthesia care unit. If the patient is transported to the intensive care unit after surgery, not the post-anesthesia care unit, then the strategy is applied until the end of surgery.
  Interventions: Other: Conventional perioperative blood pressure management strategy

INTERVENTIONS:
Other: Individualized perioperative blood pressure management strategy — In this group, perioperative mean arterial pressure and systolic blood pressure are maintained at no less than -20% of the baseline values of each patient.
  Arms: Individualized strategy
Other: Conventional perioperative blood pressure management strategy — In this group, perioperative mean arterial pressure and systolic blood pressure are maintained at ≥65 mmHg and ≥90 mmHg, respectively, in all patients.
  Arms: Conventional strategy

SUMMARY:
Study objective: To compare the effect of different perioperative blood pressure management strategies on major postoperative adverse outcomes / Study design: a multicenter, randomized controlled trial / Participants: 1896 patients undergoing major non-cardiac surgery / Methods: Patients are randomized into two groups, the individualized strategy (maintaining perioperative mean arterial pressure and systolic blood pressure more than -20% of their baseline values) or the conventional strategy (maintaining perioperative mean arterial pressure ≥65 mmHg and systolic blood pressure ≥90 mmHg in all patients). Then, the frequency of major postoperative adverse outcomes occurring within 7 postoperative days or before discharge (whichever occurs first). / Primary outcome: a composite of all-cause death, stroke, myocardial infarction, new or worsening congestive heart failure, unplanned coronary revascularization, and acute kidney injury, occuring within 7 postoperative days or before discharge (whichever occurs first).

DETAILED DESCRIPTION:
This study, aiming to reflect real clinical scenarios as much as possible, does not impose specific restrictions on perioperative management other than the target blood pressure. It allows discretion to each participating institution or physician. For the same reason, there are no restrictions on method for blood pressure measurement (invasive, non-invasive, or both), site of blood pressure measurement, fluid therapy, and vasopressors use for maintaining target blood pressure in each group.

Through random allocation, the conventional group targets a mean arterial pressure (MAP) of 65 mmHg or higher and a systolic blood pressure (SBP) of 90 mmHg or higher during surgery. The individualized group targets no less than a -20% of the baseline MAP and SBP. The baseline MAP and SBP are defined as the average values of all MAP and SBP measured between one day before surgery and the morning of the surgery.

The two blood pressure management strategies are applied until discharge from the post-anesthesia care unit. If the patient is transported to the intensive care unit after surgery, not the post-anesthesia care unit, then the blood pressure management strategies are applied until the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65 or,
* those aged ≥45 with a history of coronary artery disease, peripheral vascular disease, transient ischemic attack/stroke, or congestive heart failure,
* undergoing non-cardiac surgery under general anesthesia with an anticipated duration of ≥2 hours.

Exclusion Criteria:

* Emergency surgery
* Organ transplantation surgery
* Brain/carotid artery surgery
* American Society of Anesthesiologists physical status 5 or 6
* Pregnancy
* Uncontrolled preoperative hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg)
* Estimated glomerular filtration rate <30 ml/min/1.73m2
* Renal replacement therapy
* Acute decompensated heart failure
* Sepsis
* Shock
* Use of inotropes/vasopressor infusion (dopamine, norepinephrine, vasopressin, etc.)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1896 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative major adverse cardiac, cerebrovascular, and renal event | Occuring until discharge or postoperative day 7, whichever occurs first
  A composite of all-cause death, stroke, myocardial infarction, new or worsening congestive heart failure, unplanned coronary revascularization, and acute kidney injury.

SECONDARY OUTCOMES:
all-cause death | until discharge or postoperative day 7, whichever occurs first
  death of any cause after surgery
stroke | until discharge or postoperative day 7, whichever occurs first
  a new ischemic or hemorrhagic cerebrovascular accident with a neurological deficit confirmed by brain imaging
myocardial infarction | until discharge or postoperative day 7, whichever occurs first
  Diagnosed based on the Fourth Universal Definition of Myocardial Infarction (Type 1,2, and 3).
new or worsening congestive heart failure | until discharge or postoperative day 7, whichever occurs first
  Congestive heart failure: diagnosis on discharge letter or progression notes (medical records: pulmonary edema, congestive heart failure, etc.)
unplanned coronary revascularization | until discharge or postoperative day 7, whichever occurs first
  percutaneous coronary intervention or bypass grafting, which was not an a priori planned stepwise procedure.
acute kidney injury | until discharge or postoperative day 7, whichever occurs first
  Defined based on the serum creatinine criteria of the Kidney Disease: Improving Global Outcomes (KDIGO).
  A. Increase in serum creatinine level by 0.3 mg/dl or more within 48 hours, or B. Increase in serum creatinine level to 1.5 times the baseline or more within 7 days.
  The baseline serum creatinine level was defined as the most recent value measured prior to surgery.
Length of postoperative hospital stay (days) | assessed from the end of surgery to hospital discharge (through study completion, generally of under one month)
  Length of postoperative hospital stay described in days
Unplanned ICU admission | assessed from the end of surgery to hospital discharge (through study completion, generally of under one month)
  Unplanned intensive care unit admission after surgery
new-onset atrial fibrillation | until discharge or postoperative day 7, whichever occurs first
  New-onset atrial fibrillation of any duration captured on 12-lead electrocardiogram, continuous electrocardiogram monitoring, or telemetry.

CONTACTS AND LOCATIONS:
Overall Officials: Karam nam, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung J, Koo CH, Park J, Kim HB, Bae J, Ju JW, Lee S, Oh AR, Kim HS, Park SJ, Jeon Y, Nam K; Seoul PeRioperative OUTcome research-4 (SPROUT-4) Investigators. Effect of individualized versus conventional perioperative blood pressure management on postoperative major complications in high-risk patients undergoing noncardiac surgery: study protocol for the SPROUT-4 multicenter randomized controlled trial. Trials. 2024 Dec 26;25(1):850. doi: 10.1186/s13063-024-08707-4. PMID 39725988